CLINICAL TRIAL: NCT01452789
Title: A Randomized, Active-Control, Double-Blind, Double-Dummy Clinical Trial Comparing Sublingual Buprenorphine And Morphine Solution For The Treatment Of Neonatal Opioid Abstinence Syndrome
Brief Title: Blinded Trial of Buprenorphine or Morphine in the Treatment of the Neonatal Abstinence Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11F.193; R01DA029076-01A1 (NIH)
Record Dates: First submitted 2011-10-04; First posted 2011-10-17 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: neonatal abstinence syndrome; buprenorphine; morphine; pharmacokinetics
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Buprenorphine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sublingual buprenorphine (Experimental): This is the group that received active sublingual buprenorphine and placebo for oral morphine
  Interventions: Drug: sublingual buprenorphine
- oral morphine (Active Comparator): This is the group that received active oral morphine and placebo for sublingual buprenorphine
  Interventions: Drug: oral morphine

INTERVENTIONS:
Drug: sublingual buprenorphine — Initial daily dose: 15.9 mcg/kg/day; Initial unit dose: 5.3 mcg/kg q8 hours; Maximum daily dose: 60 mcg/kg/day; Up-titration rate: 25%; Weaning rate: 10%; Cessation Dose: Within 10 or 20% of starting dose
  Other Names: Buprenex
  Arms: sublingual buprenorphine
Drug: oral morphine — Initial daily dose: 0.4 mg/kg/day; Initial unit dose: 0.07 mg/kg q 4 hours; Maximum daily dose: 1.25 mg/kg/day; Up-titration rate: 20%; Weaning rate: 10%; Cessation Dose: 0.025 mg/kg q 4 hours
  Arms: oral morphine

SUMMARY:
The opioid neonatal abstinence syndrome (NAS) is a condition of withdrawal symptoms after utero exposure to opioids. In an open label Phase 1 trial sublingual buprenorphine was associated with a ~30% reduction length of treatment compared to standard of care morphine. Due to the subjective nature of the scoring instrument, efficacy in a blinded trial is needed to unequivocally establish the superiority of buprenorphine over morphine. The primary objective of the trial is to compare length of treatment using sublingual buprenorphine or oral morphine solution in the pharmacologic treatment of the NAS.

DETAILED DESCRIPTION:
This was a single-site, randomized, double-blind, double-dummy, parallel-group clinical trial. Potential patients were identified in the pre-natal period by staff of the Thomas Jefferson University Family center. Mothers who provided consent were contacted upon admission to TJUH. Inclusion and exclusion criteria were reassessed during the peri-partum period and study details reviewed again with the mother, and where possible, the father of the child. Women admitted to TJUH with in utero exposure to opioids who are not in the Family Center present were screened and approached for consent during their inpatient stay.

Infants at risk for NAS had abstinence assessed using the MOTHER scoring instrument, which is based upon Finnegan Score and will hereafter be called the "NAS score". This is the standard instrument used at TJUH. A need for initiation of treatment was defined as any consecutive 3 scores adding up to ≥ 24 or any single score ≥12, and the clinical decision of the attending physician that the infant requires pharmacologic therapy. Randomization took place following reaching of the threshold for initiation of treatment and a re-review of inclusion and exclusion criteria. Patients were randomized to treatment groups of 1) oral morphine/sublingual placebo for buprenorphine or 2) oral placebo for morphine/sublingual buprenorphine. Randomization was stratified according to in utero exposure to methadone or buprenorphine. Oral morphine or placebo for morphine was administered by mouth every 4 hours, while buprenorphine or placebo for buprenorphine was administered every 8 hours. NAS scores were obtained every 4 hours. Dose assessment took place on a daily basis. If the three previous NAS scores are greater than 24, a dose advancement took place (at the discretion of the neonatologist). Morphine/placebo will be increased by 20% and buprenorphine/placebo will be increased by 25%. NNNS scoring took place for all infants who provide consent at day 2-3 of life, or earlier if pharmacologic treatment is required before this time, on day 10 of life, and in the post therapy period (but no later than corrected post gestational age of 46 weeks).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 37 weeks gestation
* Exposure to opiates in utero
* Demonstration of signs and symptoms of neonatal abstinence syndrome requiring treatment

Exclusion Criteria:

* Major congenital malformations and/or intrauterine growth retardation
* Medical illness requiring intensification of medical therapy. This includes, but is not limited to suspected sepsis requiring antibiotic therapy.
* Hypoglycemia requiring treatment with intravenous dextrose.
* Bilirubin >20 mg/dL (The need for phototherapy is not exclusionary)
* Concomitant benzodiazepine or severe alcohol abuse , self-report of regular use of alcohol or of benzodiazepines use in the past 30 days, and/or receipt of benzodiazepines by prescription (as determined by self-report or intake urine) by the mother 30 days prior to birth,
* Concomitant use of Cytrochrom (CYP) 3A inhibitors (erythromycin, clarithromycin, ketoconazole, itraconazole, HIV protease inhibitors) or inducers (rifampin, carbamazepine, phenobarbital) prior to initiation of NAS treatment
* Seizure activity or other neurologic abnormality
* Breast feeding
* Inability of mother to give informed consent due to co-morbid psychiatric diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter K Kraft, MD, Principal Investigator — Thomas Jeffeson University
Locations (1):
- Thomas Jefferson University Hosptial, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Interested investigators should contact the PI listed on clinicaltrials.gov. Study protocol, statistical action plan and informed consent are available in the public domain as a supplement to the publication https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5662132/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available after Jan. 1, 2020
Access Criteria: PI and co-investigators will have discretion to share data with potential collaborators.

REFERENCES:
- [Background] Kraft WK, Dysart K, Greenspan JS, Gibson E, Kaltenbach K, Ehrlich ME. Revised dose schema of sublingual buprenorphine in the treatment of the neonatal opioid abstinence syndrome. Addiction. 2011 Mar;106(3):574-80. doi: 10.1111/j.1360-0443.2010.03170.x. Epub 2010 Oct 6. PMID 20925688
- [Background] Kraft WK, Gibson E, Dysart K, Damle VS, Larusso JL, Greenspan JS, Moody DE, Kaltenbach K, Ehrlich ME. Sublingual buprenorphine for treatment of neonatal abstinence syndrome: a randomized trial. Pediatrics. 2008 Sep;122(3):e601-7. doi: 10.1542/peds.2008-0571. Epub 2008 Aug 11. PMID 18694901
- [Derived] Zankl A, Martin J, Davey JG, Osborn DA. Opioid treatment for opioid withdrawal in newborn infants. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD002059. doi: 10.1002/14651858.CD002059.pub4. PMID 34231914
- [Derived] Kraft WK, Adeniyi-Jones SC, Chervoneva I, Greenspan JS, Abatemarco D, Kaltenbach K, Ehrlich ME. Buprenorphine for the Treatment of the Neonatal Abstinence Syndrome. N Engl J Med. 2017 Jun 15;376(24):2341-2348. doi: 10.1056/NEJMoa1614835. Epub 2017 May 4. PMID 28468518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From November 1, 2011, to May 29, 2016, we enrolled term infants (≥37 weeks of gestation) who had been exposed to opioids in utero and had signs and symptoms of the neonatal abstinence syndrome.
Period: Overall Study
Arm/Group | Sublingual Buprenorphine | Oral Morphine
Started | 33 | 30
Completed | 30 | 28
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sublingual Buprenorphine | Oral Morphine | Total
Number analyzed (Participants) | 33 | 30 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33 | 30 | 63
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: gestational age months] | 38.5 [37 to 42] | 39 [37 to 41] | 38.7 [37 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 17 | 18 | 35
Region of Enrollment [Number; unit: participants]
  United States | 33 | 30 | 63

OUTCOME MEASURES:

1. Primary Outcome: Length of Treatment
Description: This endpoint will compare length of treatment (in days) using sublingual buprenorphine or oral morphine solution.
Time Frame: Patients will be followed for the duration of hospital stay, an expected average of 5 weeks.
Population: Intention to treat
Measure: Median (Full Range); unit: days
Arm/Group | Sublingual Buprenorphine | Oral Morphine
Number analyzed (Participants) | 33 | 30
days | 15 [3 to 67] | 28 [13 to 67]
Statistical Analysis 1: Comparison: Oral Morphine; Test type: Superiority; p < 0.05, van Elteren

2. Secondary Outcome: Length of Hospitalization
Description: This endpoint will compare length of stay in the hospital (in days) using sublingual buprenorphine or morphine solution.
Time Frame: Duration of hospital stay is an expected average of 5 weeks.
Population: Intention to treat
Measure: Median (Full Range); unit: days
Arm/Group | Sublingual Buprenorphine | Oral Morphine
Number analyzed (Participants) | 33 | 30
days | 21 [7 to 71] | 33 [18 to 70]
Statistical Analysis 1: Comparison: Oral Morphine; Test type: Superiority; p < 0.05, van Elteren

3. Secondary Outcome: Number of Patients Requiring Supplemental Phenobarbital Treatment.
Description: This endpoint will compare requirement number of patients who require use of supplemental phenobarbital.
Time Frame: Patients will be followed for the duration of hospital stay, an expected average of 5 weeks.
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Sublingual Buprenorphine | Oral Morphine
Number analyzed (Participants) | 33 | 30
participants | 5 | 7
Statistical Analysis 1: Comparison: Oral Morphine; Test type: Superiority; p < 0.05, Cochran-Mantel-Haenszel

4. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Adverse events will be collected, graded by severity, and assessed for causality referent to study drug.
Time Frame: Patients will be followed for the duration of hospital stay, an expected average of 5 weeks.
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Sublingual Buprenorphine | Oral Morphine
Number analyzed (Participants) | 33 | 30
Participants | 7 | 8

ADVERSE EVENTS:
Time Frame: Adverse events were collected from allocation through discharge from hospital, up to a maximum of 71 days
Arm/Group | Sublingual Buprenorphine | Oral Morphine
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/33 | 1/30
Other Adverse Events (participants affected / at risk) | 13/33 | 10/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sublingual Buprenorphine (N=33) | Oral Morphine (N=30)
supraglottoplasty (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Associated with Pierre Robin syndrome
Inguinal hernia repair (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sublingual Buprenorphine (N=33) | Oral Morphine (N=30)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
diaper rash (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (3) — Eczematous, acneiform or vesicular; paronychia
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Umbilical granuloma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Infection (Infections and infestations) | 0 (0) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 3 (3) | 2 (3) — abdominal distension, oral thrush, allergic colitis, laryngomalacia, gastrointestinal reflux, gastrostomy tube placement

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No